CLINICAL TRIAL: NCT01193803
Title: Interest of Molecular Biology for Diagnostic of Osteo-arthritis Infections. EE Observational Prospective Study
Brief Title: Molecular Microbiology in Osteo-arthritis Infection
Acronym: MOLOS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRC076057; 297-08 (Other: CEERB)
Record Dates: First submitted 2010-04-01; First posted 2010-09-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Osteoarticular Infections
Keywords: Prosthetic Joint Infections; Vertebral Osteomyelitis; Septic arthritis; Molecular methods
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Detection of bacteria will be performed on sample provided from the osteoarticular infections like articular fluids, synovial biopsies, bone biopsies, intervertebral disc, paravertebral or epidural abscess, articular capsul...
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Spondylodiscitis control group: Patients needing vertebral biopsy looking for tumoral etiology
  Interventions: Procedure: Microbiological cultures and Molecular biology
- Prosthetic Joint Infection control group: Patients with primary prosthetic arthrosis surgery
  Interventions: Procedure: Microbiological cultures and Molecular biology
- Septic arthritis control group: Arthrosic patients needing evacuating articular punction with leucocytes infiltration less than 1000 /mm3
  Interventions: Procedure: Microbiological cultures and Molecular biology
- Spondylodiscitis case group: Patients suspected of Discitis and/or Vertebral Osteomyelitis is defined by the need of spinal biopsy in infectious context.
  Interventions: Procedure: Microbiological cultures and Molecular biology
- Prosthetic Joint Infection case group: Patients suspected of Prosthetic Joint Infection defined by the need of surgical revision for diagnostic or therapeutic aiming in infectious context.
  Interventions: Procedure: Microbiological cultures and Molecular biology
- Septic arthritis case group: Patients suspected of Septic arthritis without prosthesis were defined by the need of synovial punction and/or biopsy
  Interventions: Procedure: Microbiological cultures and Molecular biology

INTERVENTIONS:
Procedure: Microbiological cultures and Molecular biology — Biological/Vaccine: Microbiological cultures and Molecular Biology Bacteriological procedures: All solid specimens will be crushed using a mechanic apparatus. Direct examination and cultures will be performed according to the guidelines applied for osteoarticular infections. Cultures and subcultures will be incubated for 15 days to 3 months for Mycobacteria.
  Molecular procedures: DNA extraction will be based on Boom's method (QIAGEN kit and EZ1 BioRobot). Detections of bacteria will be performed by amplification and sequencing of the 16S rRNA gene. Some specific detections as the detection of Staphylococcus sp. and Mycobacterium tuberculosis will be added to this protocol.

SUMMARY:
Osteoarticular infections are painful and disabling diseases that require antimicrobial treatment adapted to the microorganisms implicated. Microbiological cultures are currently regarded as the reference for identification of pathogenic bacteria. However, the sensitivity of these cultures is very variable and depends both on the context in which clinical samples are taken, and on the pathogen involved. The rate of detection varies according to infection type: from 50 to 70% for infectious spondylodiscitis, 65 to 95% for prosthetic joint infections, 50% for gonococcal arthritis and 90% for non-gonococcal arthritis. The aim of the study is to evaluate the diagnostic performances of microbiological cultures and molecular methods in case of osteoarticular infections. The gold standard will be established by an expert group of osteoarticular infection (composed by a bacteriologist, a radiologist, a surgeon, an anatomy-pathologist and a rheumatologist), which established the final diagnosis of infected or not infected patients.

DETAILED DESCRIPTION:
Background: Osteoarticular infections are painful and disabling diseases that require antimicrobial treatment adapted to the microorganisms implicated. Microbiological cultures are currently regarded as the reference for identification of pathogenic bacteria and it seems that the microbiological cultures are sufficient in most cases to establish the diagnosis. However, the sensitivity of these cultures is very variable and depends both on the context in which clinical samples are taken, and on the pathogen involved. In addition, previous experimental data show that molecular methods could produce a diagnosis missing by conventional cultures. Main objective: The aim of the study is to evaluate the diagnostic performances of microbiological cultures and molecular method by considering for the definition of cases an accumulation of clinical, radiological and biological arguments usually used to establish the diagnosis of bone and joint infections. The discordance of the two methods will be secondary classified by an expert group of osteoarticular infection (composed by a bacteriologist, a radiologist, a surgeon, a anatomy-pathologist and a rheumatologist).Tested hypothesis:Interest of molecular methods for the diagnosis of osteoarticular infections.Secondary objective:Quantification of the delay of the results obtained by the two methods Study design: · One centre specialized in osteoarticular infections· Observational prospective study· Two methods of diagnosis: cultures and molecular methods· An expert group Included patients and number of patients: Total of 284 patients composed by 194 cases and 90 controlsIncluded patients (n=194) will all have a suspected diagnosis of osteoarticular infections included discitis, septic arthritis and prosthetic joint infection defined by inclusions criteria.Results of the included patients will be compared to those obtained from the group of control patients (n=90).Protocol of duration: Study duration is 6 months for each patientThe protocol duration is planned for 2 yearsProcedures:All samples will be treated with the same procedure - Samples (synovial fluids, biopsies, ..) will be recovered either during surgery, by puncture aspiration at the bedside, or by guided ultrasonography, all under sterile conditions (mask, sterile gloves, cautious skin preparation and towelling) and transported to the Bacteriology department in sterile tubes without additional substrate in less than 12 hours. - Bacteriological procedures will be performed according to the guidelines applied for osteoarticular infection · Liquid samples: erythrocyte and leukocyte counts, polymorphonuclear percentage · Solid specimens: crushed using a mechanic apparatus · Gram and auramine staining· Cultures at 37°C on Columbia sheep blood agar (aerobically and anaerobically for 5 days), chocolate agar supplemented with IsoVitaleX (with 5% CO2 for 5 days), brain heart infusion broth (anaerobically for 15 days with subcultures done after 10 days on the same agar media, even if aspect was not cloudy).· Mycobacterial culture : Lowenstein-Jensen and COLETSOS media, MGIT incubated for 3 months.- Molecular procedures· DNA manipulations pre- and post-PCR: in separate rooms with separate pipetting devices to prevent contamination of samples with foreign DNA. · Equipment used in pre-PCR steps: DNA-free and UV-irradiated. · DNA extraction based on Boom's method: QIAGEN kit and EZ1 BioRobot · Broad-range 16S rRNA gene amplification · Amplicons: sequenced in both directions on an ABIPRISM 3100 analyser (Applied Bio systems, COURTABOEUF, France). · Cloning experiments for several sequences in one sample· Analysis of sequence: GenBank using the BLASTN program through the website of the National Centre of Biotechnology Information.· Internal control PCR: b-actin gene· Real time PCR: for the detection of mycobacteria and gonococcal arthritis- Potential implications: We could have chosen, like the majority of the studies published to date, to compare our molecular method with another method of diagnosis (culture, histology). However, there is not currently gold standard and the diagnosis of osteoarticular infections generally rests on an accumulation of arguments. The rule of the expert group is to determine, with less possible error, if each patient included will be "infected". This methodology is close to daily clinical reality and trusted in physician who was treating the patient. If the study shows an advantage of the molecular biology versus classical methods in our groups it would then be justified to discuss the diagnosis diagram of osteoarticular infections.

ELIGIBILITY:
Inclusion Criteria:

* Patient are more than 18 years old
* Patient who do not declined to have his medical records reviewed for research

Spondylodiscitis (S) group:

* Patients suspected of Discitis and/or Vertebral Osteomyelitis is defined by the need of spinal biopsy in infectious context. Spinal biopsies will be justified by one or more clinical or imaging findings:
* Clinical presentation
* Spinal pain unrelieved by rest
* Localized tenderness, Neurological deficits or limited range of motion
* Fever > 38°C

  * Imaging findings (plain radiographs, MRI or CT):
* Erosions of end plates on adjacent vertebral bodies
* Decreased height of the intervertebral disk
* Presence of a nonvascularized zone suggesting presence of pus or necroses in intervertebral, epidural space or in paraspinal soft-tissues

Prosthetic Joint Infection (PJI) Group

Patients suspected of Prosthetic Joint Infection were defined by the need of surgical revision for diagnostic or therapeutic aiming in infectious context. This revision will be justified by one or more clinical, biological or imaging findings:

Clinical presentation

* Persistent joint pain
* Fever > 38°C
* Erythematous, swollen, fluctuant, and/or tender surgical wound
* Wound dehiscence
* Limited range of joint motion

Biological findings

* CRP > 10 mg/l
* Synovial leukocytes count > 1500/mm3 and polymorphonuclear leukocytes > 65%

Imaging findings

* Prosthesis loosening: Periprosthetic osteolysis, progressive peri-prosthetic edging
* Scintigraphy by means of a technetium (Tc99m) scan, gallium citrate (Ga67) scan, or indium (In111)-labeled leukocyte showing fixation around the prosthesis.

Septic arthritis (SA) Group

* Patients suspected of Septic arthritis without prosthesis were defined by the need of synovial punction and/or biopsy justified by one or more clinical, biological or imaging findings:

Clinical presentation

* Acute joint pain and/or swelling
* Adenopathy near inflammatory joint
* Fever > 38°CBiological findings
* WBC > 10 000/ mm3
* CRP > 10 mg/l
* Synovial leukocytes count > 2000/mm3 or polymorphonuclear leukocytes > 90%

Imaging findings:

* Capsular and surrounding soft-tissues swelling
* Synovial notch and/or demineralization
* Periarticular Abscess

Exclusion criteria:

* Patients already include.
* Patient without health insurance
* Antibiotic treatment before sampling does not constitute an exclusion criterion

Exclusion criteria for control groups:

Patient with one or more criteria:

* Suspicion of concomitant infection defined by a fever >38°C and CRP > 10mg/l
* Arthrosis treated by infiltration in the 6 months which preceding inclusion
* Rapidly progressive arthrosis Prosthesis loosening or bone necrosis presumed to be aseptic
* Patients with prior spinal instrumentation or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected diagnosis of osteoarticular infections included discitis, septic arthritis and prosthetic joint infection and control patients.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prosthetic Joint Infections, Vertebral Osteomyelitis and Septic arthritis: Frequency of detection with classical bacteriological methods and molecular methods | Day 0

SECONDARY OUTCOMES:
Time of returned results by one or the other of the techniques | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice BERCOT, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital LARIBOISIERE, Paris, France

REFERENCES:
- [Background] Fihman V, Hannouche D, Bousson V, Bardin T, Liote F, Raskine L, Riahi J, Sanson-Le Pors MJ, Bercot B. Improved diagnosis specificity in bone and joint infections using molecular techniques. J Infect. 2007 Dec;55(6):510-7. doi: 10.1016/j.jinf.2007.09.001. Epub 2007 Oct 29. PMID 18029022